CLINICAL TRIAL: NCT01776138
Title: PORCH: A Registry of Prospective Outcomes of Radical Cystectomy With or Without Chemotherapy
Brief Title: Study of Outcomes After Surgery/Treatment to Treat Bladder Cancer
Acronym: PORCH
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1206; 12-0577 (Other: UNC IRB)
Record Dates: First submitted 2012-09-20; First posted 2013-01-25 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Bladder Cancer
Keywords: Elderly; Chemotherapy; Cystectomy; Radical Cystectomy; University of North Carolina; Cancer; Bladder Cancer; Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms | interventions — Surveys and Questionnaires; Geriatric Assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bladder Cancer Patients: Patients diagnoses with bladder cancer who are eligible to undergo treatment.
  Interventions: Other: Collect Blood and Survey Instruments

INTERVENTIONS:
Other: Collect Blood and Survey Instruments
  Other Names: p16 Blood Collection; Geriatric Assessment; Fact-BL; Health Behavior Questionnaire

SUMMARY:
The purpose of this study is to create a registry of older patients undergoing surgical and/or medical treatment for bladder cancer. The registry will record side-effect and outcomes related to the treatment using different surveys and biological measures.

DETAILED DESCRIPTION:
The primary purpose of this protocol is to create a registry of elderly patients with high-risk invasive bladder cancer undergoing radical cystectomy with or without preoperative chemotherapy.

Secondary objectives will include an exploration of the association between functional status, surgical complications, and laboratory markers with complications and survival. In addition, exploratory analyses may evaluate the association of expression of the senescence marker p16INK4a and the morbidity and mortality associated with treatment.

Patients will be asked to complete a Geriatric Assessment (GA) and FACT-Bl serially over the course of the study in order to evaluate their functional status and quality of life during the course of treatment. Additionally, complications will be tracked in an inpatient and outpatient setting using the Memorial Sloan Kettering Cancer Center (MSKCC) complications grading system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a known pathologic diagnosis of lower tract urothelial carcinoma who are eligible to undergo radical cystectomy with or without neoadjuvant chemotherapy for definitive diagnosis and treatment.
* Signed, IRB approved written informed consent.
* Completion of baseline Geriatric Assessment

Exclusion Criteria:

* Inability to read and speak English
* Inability to comply with study for any other reason than language
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a known pathologic diagnosis of lower tract urothelial carcinoma who are eligible to undergo radical cystectomy with or without neoadjuvant chemotherapy for definitive diagnosis and treatment.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2012-07-23 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
To collect the number of changes in functional status, surgical complications and survival status collected in a prospective database of patients undergoing a radical cystectomy with or without chemotherapy | 1 Year
  To collect the number of changes in functional status, surgical complications, and survival in patients with urothelial carcinoma of the bladder following radical cystectomy with or without neoadjuvant chemotherapy in a prospective database (to be called the PORCH database- "Prospective Outcomes of Radical cystectomy with or without Chemotherapy").

SECONDARY OUTCOMES:
To measure associations between baseline measures with post-surgery and 90 day outcome measures | 2 years
  Measure the association of all baseline measures with the outcomes of complications post-surgery and 90 day mortality for the 25 patients entered into the database who complete the GA and FACT-Bl questionnaires.
To count changes over the course of treatment for components of the GA, the FACT-Bl, p16, and other clinical characteristics. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela Smith, MD, Principal Investigator — University of North Carolina Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States